CLINICAL TRIAL: NCT07290868
Title: Scaling up Personalized mHealth-supported Resistance Training and Education for Children and Adolescents With Type 1 Diabetes: The Diactive-1 v2.0 Randomized Controlled Trial
Brief Title: Diactive-1: Scaled-up Personalized mHealth Program for Youth With Type 1 Diabetes
Acronym: Diactive-1v2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Universidad Pública de Navarra (Other); University of Valencia (Other); Instituto de Investigación Sanitaria de Navarra (IdiSNA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGH_Diactive1_2025
Record Dates: First submitted 2025-12-15; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: mHealth; Resistance training; Education; Handgrip strength
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diactive-1 (Experimental): The intervention in the experimental group will center around the use of a mobile application (i.e., device), namely the Diactive-1 app.
  Interventions: Device: Diactive-1
- Waiting-list control group (No Intervention): This arm will not complete an intervention. Participants will be instructed to continue to follow their normal daily diabetes care plan (i.e., standard care). This group will be granted access to the app following the intervention.

INTERVENTIONS:
Device: Diactive-1 — Participants will engage in a 12-week resistance exercise program with the goal of maintaining at least 3 sessions per week, with 3-6 exercises per session (≈13-33 minutes). Participants will be able to choose among three training formats, traditional resistance training, Tabata/high-intensity intervals, or circuit training, and may perform the sessions individually or in pairs, depending on preference and feasibility at the center. The training intervention will comprise 3-4 sets of 6-12 repetitions and will consist of a combination of exercises for the upper body, lower body, and core, using primarily the participants' own body weight. The load and intensity of the exercise will be adjusted according to the number of repetitions and the difficulty/progression of the selected exercises. A mobile application (Diactive-1) will be used to deliver, monitor, and record the sessions.
  Arms: Diactive-1

SUMMARY:
The Diactive-1 project aims to establish the Diactive-1 mobile application as a clinical tool for managing type 1 diabetes in children and adolescents in several hospitals from Spain. The successful implementation of the app in new healthcare centers nationwide represents a key step toward the development of a comprehensive and scalable program. This approach seeks not only to optimize current patient care but also to democratize access to an innovative, evidence-based intervention that supports daily diabetes management.

In this new phase, the project will integrate the application into routine clinical care for patients with type 1 diabetes through the use of a simple handgrip strength measurement. A dedicated web platform (www.diactive.es) is being developed to allow clinicians to enter basic patient data, including handgrip strength, sex, and email address. Based on this information, the system will automatically generate a personalized download link for the Diactive-1 app, accompanied by tailored guidance and an initial fitness level classification (low, medium, or high) according to European reference values.

This process will define each user's baseline fitness level and facilitate the use of Diactive-1 as an integrated and individualized disease management tool. The ultimate goal is to strengthen clinical decision-making, improve patient engagement, and extend the benefits of digital health to a broader pediatric population living with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 Diabetes Mellitus (T1DM) for 6 months or longer (requiring >0.5 U/kg/day of insulin and having HbA1c >6%, i.e., not in the "honeymoon phase").
* Receiving multiple daily injection (MDI) therapy or insulin pump therapy (CSII).
* Signed informed consent authorizing legal participation in the research project (child/adolescent and parent(s)/legal guardian).
* Availability to participate in the study using an m-Health application (Diactive-1) designed for the programming of muscle-bone strengthening physical exercise.
* Understanding of Spanish.

Exclusion Criteria:

* Comorbidities that limit the ability to engage in physical activity.
* Lack of internet access when using the application, whether due to Wi-Fi, mobile data, or international roaming issues.
* Absence of a mobile phone or tablet with an Android or iOS (Apple) operating system, or no family member willing to lend a device for each session using the application for study-related purposes.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in handgrip strength | Baseline and 12 weeks
  Handgrip strength measured in kilograms using the Takei III Smedley Type Digital Dynamometer

SECONDARY OUTCOMES:
Change in daily insulin dose requirement | Baseline and 12 weeks
  The daily insulin dose requirements will be measured in units per kilogram of body weight. Assessment will rely on participant-reported data from insulin pumps or injection logs, gathered for 7 days prior to the intervention and after the intervention.
Change in glycated hemoglobin | Baseline and 12 weeks
  Glycated hemoglobin (measured in percent)
Number of participants with good glycemic control | Baseline and 12 weeks
  Number of participants with a glycated hemoglobin level lower than 7%
Change in time in range | Baseline and 12 weeks
  The percentage of time a person spends with their blood glucose levels in the target range (70-180 mg/dL or 3.9-10 mmol/L) (measured in percent)
Change in time below range | Baseline and 12 weeks
  The percentage of time a person spends with their blood glucose levels below the target range (<70 mg/dL or <3.9 mmol/L, i.e., hypoglycemia) (measured in percent)
Change in time above range | Baseline and 12 weeks
  The percentage of time a person spends with their blood glucose levels above the target range (>180 mg/dL or 10 mmol/L, i.e., hyperglycemia) (measured in percent).
Change in glycemic variability | Baseline and 12 weeks
  Glycemic variability measures the fluctuation in blood glucose levels over time, expressed as a percentage. Lower glycemic variability indicates more stable levels, while higher glycemic variability suggests greater fluctuations.
Change in compliance with 24-hour movement behaviors | Baseline and 12 weeks
  Physical activity at different intensities (average min/day), sedentary time (average min/day) and sleep (average min/day) will be measured using self-reported questionnaires.
Change in self-reported physical activity | Baseline and 12 weeks
  Aerobic and muscle-strengthening activities will be assessed using two separate ad hoc questions. Participants will have response options ranging from 0 to 7 days per week, with increments of 1 day.
Change in self-reported physical fitness | Baseline and 12 weeks
  The International Fitness Scale (IFIS) will be used to assess self-reported physical fitness. This scale includes five elements that will employ a 5-point Likert scale to inquire about children's overall perception of their physical fitness, as well as their perception of their cardiorespiratory fitness, muscular fitness, speed-agility, and flexibility compared to their peers. The Likert scale will provide choices ranging from 'very poor' to 'poor,' 'average,' 'good,' and 'very good' physical fitness.
Change in sleep duration | Baseline and 12 weeks
  Sleep duration will be determined by recording the number of hours slept each day
Change in physical literacy | Baseline and 12 weeks
  Physical literacy will be assessed using the Spanish Perceived Physical Literacy Instrument (S-PPLI), a 9-item questionnaire that evaluates three dimensions: knowledge and understanding; self-expression and communication; and sense of self and self-confidence
Change in physical activity barriers | Baseline and 12 weeks
  We will use the Spanish adaptation of the Physical Activity Barriers Scale for pediatric type 1 diabetes (PABS-1), a validated instrument for assessing perceived barriers to physical activity in children and adolescents with type 1 diabetes
Adherence to the Mediterranean Diet | Baseline and 12 weeks
  For assessing adherence to the Mediterranean Diet, the KIDMED index will be employed. This index provides a score on a scale of 0 to 12, with higher scores indicating stronger adherence.
Change in disordered eating | Baseline and 12 weeks
  Disordered eating will be screened using the mSCOFF questionnaire. This questionnaire consists of six straightforward yes/no questions. A positive response to two or more of these questions suggests a potential eating disorder, often requiring further evaluation.
Change in subjective well-being | Baseline and 12 weeks
  Subjective well-being will be assessed using the CUBE questionnaire, which comprises five items that evaluate different aspects of life satisfaction and emotional states.
Change in Health-Related Quality of Life | Baseline and 12 weeks
  Health-Related Quality of Life will be evaluated using the Screening for and Promotion of Health-Related Quality of Life in Children and Adolescents (KIDSCREEN-10).
Change in Health-Related Quality of Life in the context of a chronic illness | Baseline 12 weeks
  Health-Related Quality of Life in the context of a chronic illness will be evaluated using the Spanish version of the 'Questionnaire for Young People with Diabetes' (DISABKIDS).
Change in microalbuminuria | Baseline and 12 weeks
  Microalbuminuria will be evaluated as an indicator of early kidney involvement. A first-morning urine sample will be collected, and the albumin-to-creatinine ratio (ACR) will be determined using standardized laboratory procedures. Values will be expressed in mg/g. Microalbuminuria will be defined as an ACR between 30 and 300 mg/g, according to international diabetes guidelines.
Change in retinal findings | Baseline and 12 weeks
  Retinal imaging will be performed to assess early signs of diabetic retinopathy. Images of both eyes will be captured following standard ophthalmologic protocols and evaluated by trained specialists. Findings will be categorized as no retinopathy, mild, moderate, or severe diabetic retinopathy, based on international classification criteria.
Change in body mass index | Baseline and 12 weeks
  Weight and height will be combined to report body mass index in kg/m^2
App usability: user | 12 weeks
  The usability of the app will be evaluated using the Spanish Version of the User Version of the Mobile Application Rating Scale (uMARS).
App usability: expert evaluation | 12 weeks
  We will employ the Spanish adaptation of the Mobile Application Rating Scale (MARS), a standardized instrument for expert appraisal of mHealth applications.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Miguel Servet/ Navarrabiomed, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No